CLINICAL TRIAL: NCT06249542
Title: Implementing Routine Screening for Cannabis and Other Drug Use Disorders in Primary Care: Impact on Diagnosis and Treatment in a Randomized Pragmatic Trial in 22 Clinics
Brief Title: Implementing Screening for Cannabis and Other Drug Use Disorders in Primary Care: Impact on Diagnosis and Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 5R01DA047312 (NIH); 5R01DA047312 (NIH)
Record Dates: First submitted 2023-07-20; First posted 2024-02-08 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Cannabis-Related Disorder; Cannabis Abuse; Drug Abuse; Drug Use Disorders; Opioid Use Disorder; Opioid Abuse; Substance Abuse; Substance Use Disorders
MeSH Terms: conditions — Marijuana Abuse; Substance-Related Disorders; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care Delivery Improvement Intervention (Experimental): The care delivery improvement intervention consisted of a period of 4 months during which practice facilitators supported each clinic in implementing routine, population-based screening, assessment, treatment, and follow-up for depression and unhealthy substance use and substance use disorders.
  Interventions: Other: Care Delivery Improvement Intervention
- Usual Care (No Intervention): Usual care consisted of care received in a study clinic after January 1, 2015 and prior to active implementation of the quality improvement intervention in that clinic. The usual care period included 1) a two-month pre-intervention preparatory period during which EHR tools designed to support the intervention had been activated in the EHR and were available to clinic staff but had not yet been actively promoted by practice facilitators (a condition the investigators refer to as "passive access"), and 2) a two-month preparation period during which practice facilitators, who were not members of the local clinic staff, engaged clinic staff in team building exercises and pretesting of the intervention.

INTERVENTIONS:
Other: Care Delivery Improvement Intervention — KPWA clinical leaders and clinicians in each clinic implemented all aspects of the care delivery improvement intervention, including screening, assessment, and shared decision-making followed, as appropriate, by treatment. The implementation strategy, which was refined during the pilot phase, included:
  1. Identification of a clinical champion and local implementation team
  2. Participatory design
  3. Training of primary care providers and medical assistants
  4. Use of EHR clinical decision support tools
  5. Weekly facilitated local implementation team meetings
  6. Performance monitoring with feedback, including monthly meetings with the local implementation team and clinic leaders
  7. Learning sessions for primary care providers during implementation
  8. Social worker use of an EHR registry with weekly supervision
  9. Use of a video and informational handouts to shift attitudes and reduce stigma associated with unhealthy substance use
  Arms: Care Delivery Improvement Intervention

SUMMARY:
Our proposed evaluation study is designed to evaluate the impact of a recently completed stepped wedge cluster randomized trial, conducted at Kaiser Permanente Washington (KPWA), of an intervention to improve care and management of patients with drug use disorders (DUDs) in primary care (Aim 1). We will also explore the reasons for any apparent gaps in DUD care by analyzing clinicians' free-text encounter notes using manual chart review, natural language processing (NLP), and/or NLP-assisted manual chart review, as appropriate (Aim 2).

Specific Project Aims are as follows:

Aim 1 The primary research question we address in Aim 1 is whether routine screening for drug use disorders in primary care (PC) settings increases DUD treatment. We define DUDs as including opioid use disorders (OUD), cannabis use disorders (CUD), and other non-alcohol drug use disorders (OTH). Previously published analyses indicate that the 22 PC clinics in this trial sustained very high rates of screening (88%) and a 3-clinic DUD pilot study suggested that this screening resulted in increased diagnosis of CUD and increased treatment of DUDs in general, even at relatively low observed rates of PC-based screening and assessment.

Aim 2

The overall goal of Aim 2 is to expand our understanding of gaps in DUD diagnosis and treatment that persist-despite implementation of high rates of PC screening and assessment for SUDs-using rich information available only in free-text chart notes. Through analysis of relevant chart notes Aim 2 of this project will descriptively characterize gaps in DUD diagnosis and DUD treatment (i.e., instances where information in a patient's record suggests a DUD could be diagnosed but no diagnosis is present, or a new diagnosis suggest treatment is indicated but no evidence of treatment is present), and characterize reasons for DUD care gaps.

DETAILED DESCRIPTION:
Prior to 2015, KPWA's Behavioral Health Service (BHS) leaders decided to implement an intervention to improve the quality of population-based primary care of several behavioral health conditions including depression and unhealthy use of alcohol, opioids, cannabis, and other drugs. Additionally, these leaders decided to transition primary care social workers to become integrated behavioral health clinicians in 2015.

Pilot testing of quality improvement implementation strategies in 2015 was led by BHS leaders in collaboration with other KPWA departments. State-of-the-art implementation methods were used to integrate evidence-based alcohol-related care into 3 pilot primary care clinics. Implementation strategies included: participatory design, clinical champions, practice facilitation, performance monitoring and feedback, and clinical decision support in the electronic health record (EHR). To encourage care team members to routinely engage patients in discussions of unhealthy substance use while avoiding stigmatized language, a video and informational handout was designed and used in an effort to shift caregiver attitudes and practices. Screening and follow-up assessment for symptoms of all substance use disorders are conducted on paper and entered into the KPWA Epic EHR by medical assistants. The implementation strategy was refined through the use of ongoing formative evaluation.

Timing of the implementation of the quality improvement intervention was staggered to 1) allow adequate support of care teams by available care practice facilitators, and 2) facilitate rigorous evaluation of the impact on patient care of implementing the intervention using secondary quality improvement data.

Research teams at Kaiser Permanente Washington Health Research Institute (KPWHRI) supported the implementation effort and have lead or are leading various components of the evaluation. All evaluations are based on a pragmatic stepped-wedge quality improvement randomized trial design for 22 KPWA clinics. Three pairs of these clinics were combined for purposes of implementation and evaluation, resulting in a set of 19 implementation "sites." Implementation was staggered in 7 waves over a three-year period, with each wave including 2 or 3 sites (3 waves in the first year and 4 waves in each of the second and third years). Randomization was also stratified by year. For pragmatic reasons, KPWA clinical leaders designated 9 clinics that were randomized in the first year (as 9 sites). The remaining 13 clinics were randomized in the second and third years (as 10 sites).

The implementation period in each clinic lasted 4 months.

Our definitions of drug use disorder treatment are modified versions of definitions published in the Healthcare Effectiveness Data and Information Set (HEDIS).

ELIGIBILITY:
Inclusion Criteria:

* Kaiser Permanente Washington health plan enrollees, AND
* Age 18 years and older, AND
* Completes one or more encounters in any study clinic during the study period

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 363936 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Rate of new drug use disorder treatment using modified HEDIS criteria. | Between 1 and 12 months per year
  A patient has a new episode of treatment for a drug use disorder when: 1) they receive a new diagnosis (i.e., a disorder diagnosis preceded by 365 days without a diagnosis of the same type) for a specific disorder type--OUD, CUD, or OTH, 2) they initiate drug use disorder treatment, defined as evidence of a 2nd encounter coded with the same type of disorder diagnosis 1-14 days following the above defined new diagnosis, and 3) they engage in drug use disorder treatment, defined as two additional encounters coded with diagnoses of the same type of disorder 1-29 days after meeting the above treatment initiation criterion. Each patient may contributed between one month and 12 months per calendar year, including all months in which they have at least one study clinic encounter. The outcome rate is calculated per study clinic per month as the number of patients meeting this outcome definition per 10,000 patients with study clinic encounters.

SECONDARY OUTCOMES:
Rate of new diagnosis of drug use disorders, all drug types combined | Between 1 and 12 months per year
  Rates of new diagnoses of drug use disorders are defined operationally as the presence of an encounter in a study clinic coded with a drug use disorder diagnosis not preceded by an encounter during the prior 365 days in any setting coded with a drug use disorder diagnosis of the same type (i.e., OUD, CUD, or OTH).
Rate of new diagnosis of opioid use disorders | Between 1 and 12 months per year
  Rates of new diagnoses of opioid use disorders are defined operationally as the presence of an encounter in a study clinic coded with an opioid use disorder diagnosis not preceded by an encounter during the prior 365 days in any setting coded with an opioid use disorder diagnosis.
Rate of new diagnosis of cannabis use disorders | Between 1 and 12 months per year
  Rates of new diagnoses of cannabis use disorders are defined operationally as the presence of an encounter in a study clinic coded with a cannabis use disorder diagnosis not preceded by an encounter during the prior 365 days in any setting coded with a cannabis use disorder diagnosis.
Rate of new diagnosis of other drug use disorders | Between 1 and 12 months per year
  Rates of new diagnoses of other drug use disorders are defined operationally as the presence of an encounter in a study clinic coded with an other drug use disorder diagnosis (which includes disorders involving any substances other than opioids, cannabis, and alcohol) not preceded by an encounter during the prior 365 days in any setting coded with an other drug use disorder diagnosis.
Rate of opioid use disorder treatment using a modified HEDIS operational definition. | Between 1 and 12 months per year
  A patient has this outcome when: 1) they receive a new diagnosis (i.e., a disorder diagnosis preceded by 365 days without a diagnosis of the same type) for opioid use disorder, 2) they initiate opioid use disorder treatment, defined as evidence of a 2nd encounter coded with an opioid use disorder diagnosis 1-14 days following the above defined new diagnosis, and 3) they engage in opioid use disorder treatment, defined as two additional encounters coded with opioid use disorder diagnoses 1-29 days after meeting the above defined treatment initiation criterion. Each patient may contributed between one month and 12 months per calendar year, including all months in which they have at least one study clinic encounter. The outcome rate is calculated per study clinic per month as the number of patients meeting this outcome definition per 10,000 patients with study clinic encounters.
Rate of cannabis use disorder treatment using a modified HEDIS operational definition | Between 1 and 12 months per year
  A patient has this outcome when: 1) they receive a new diagnosis (i.e., a disorder diagnosis preceded by 365 days without a diagnosis of the same type) for cannabis use disorder, 2) they initiate cannabis use disorder treatment, defined as evidence of a 2nd encounter coded with a cannabis use disorder diagnosis 1-14 days following the above defined new diagnosis, and 3) they engage in cannabis use disorder treatment, defined as two additional encounters coded with cannabis use disorder diagnoses 1-29 days after meeting the above defined treatment initiation criterion. Each patient may contributed between one month and 12 months per calendar year, including all months in which they have at least one study clinic encounter. The outcome rate is calculated per study clinic per month as the number of patients meeting this outcome definition per 10,000 patients with study clinic encounters.
Rate of other drug use disorder treatment using a modified HEDIS operational definition | Between 1 and 12 months per year
  A patient has this outcome when: 1) they receive a new diagnosis for an other drug use disorder (i.e., disorders involving any substance type other than opioids, cannabis, and alcohol) preceded by 365 days without a diagnosis of the same type, 2) they initiate other drug use disorder treatment, defined as evidence of a 2nd encounter coded with an other drug use disorder diagnosis 1-14 days following the above defined new diagnosis, and 3) they engage in other drug use disorder treatment, defined as two additional encounters coded with other drug use disorder diagnoses 1-29 days after meeting the above defined treatment initiation criterion. Each patient may contributed between one month and 12 months per calendar year, including all months in which they have at least one study clinic encounter. The outcome rate is calculated per study clinic per month as the number of patients meeting this outcome definition per 10,000 patients with study clinic encounters.

CONTACTS AND LOCATIONS:
Overall Officials: David S Carrell, PhD, Principal Investigator — Kaiser Permanente

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glass JE, Bobb JF, Lee AK, Richards JE, Lapham GT, Ludman E, Achtmeyer C, Caldeiro RM, Parrish R, Williams EC, Lozano P, Bradley KA. Study protocol: a cluster-randomized trial implementing Sustained Patient-centered Alcohol-related Care (SPARC trial). Implement Sci. 2018 Aug 6;13(1):108. doi: 10.1186/s13012-018-0795-9. PMID 30081930
- [Background] Bobb JF, Lee AK, Lapham GT, Oliver M, Ludman E, Achtmeyer C, Parrish R, Caldeiro RM, Lozano P, Richards JE, Bradley KA. Evaluation of a Pilot Implementation to Integrate Alcohol-Related Care within Primary Care. Int J Environ Res Public Health. 2017 Sep 8;14(9):1030. doi: 10.3390/ijerph14091030. PMID 28885557